CLINICAL TRIAL: NCT01499082
Title: 6-Month, Multicenter, Randomized, Open-label, Parallel-group Study Comparing the Efficacy and Safety of a New Formulation of Insulin Glargine and Lantus® Both Plus Mealtime Insulin in Patients With Type 2 Diabetes Mellitus With a 6-month Safety Extension Period
Brief Title: Comparison of a New Formulation of Insulin Glargine With Lantus in Patients With Type 2 Diabetes Mellitus on Basal Plus Mealtime Insulin
Acronym: EDITION I
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EFC11628; 2010-023769-23 (EudraCT Number)
Record Dates: First submitted 2011-12-16; First posted 2011-12-26 (Estimated); Results first posted 2015-04-23 (Estimated); Last update posted 2022-03-25 (Actual); Status verified 2022-03

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Glargine

ARMS (2):
- HOE901-U300 (Experimental)
  Interventions: Drug: HOE901-U300 (new formulation of insulin glargine)
- Lantus (Active Comparator)
  Interventions: Drug: Lantus (insulin glargine)

INTERVENTIONS:
Drug: HOE901-U300 (new formulation of insulin glargine) — HOE901-U300 (new insulin glargine 300 units per milliliter [U/mL]) subcutaneous (SC) injection once daily (evening) for 12 months on top of mealtime insulin analogue. Dose titration seeking fasting plasma glucose 4.4-5.6 millimole per liter (mmol/L) (80 - 100 milligram per deciliter [mg/dL]). After 6 months participants were proposed to participate to the administration substudy and to receive either HOE901-U300 once daily at intervals of 24 +/- 3 hours (adaptable dosing intervals) or to continue once daily injections of HOE901-U300 every 24 hours (fixed dosing intervals) up to Month 9.
  Arms: HOE901-U300
Drug: Lantus (insulin glargine) — Lantus (HOE901-U100, insulin glargine 100 U/mL) SC injection once daily (evening) for 12 months on top of mealtime insulin analogue. Dose titration seeking fasting plasma glucose 4.4-5.6 mmol/L (80 - 100 mg/dL).
  Other Names: Lantus
  Arms: Lantus

SUMMARY:
Primary Objective:

* To compare the efficacy of insulin glargine new formulation and Lantus in terms of change in HbA1c from baseline to endpoint (scheduled month 6) in adult participants with type 2 diabetes mellitus

Secondary Objectives:

* To compare the efficacy of insulin glargine new formulation and Lantus in terms of occurrence of nocturnal Hypoglycemia

DETAILED DESCRIPTION:
The maximum study duration was up to approximately 58 weeks per participant, consisting of:

* up to 2 week screening period
* 6-month comparative efficacy and safety treatment period
* 6-month comparative safety extension period
* 4-week safety follow-up period in a subset of participants
* a 3-month administration substudy period starting after completion of the 6-month study period for participants willing to in a subset of participants randomized to HOE901-U300

ELIGIBILITY:
Inclusion criteria :

* Participants with type 2 diabetes mellitus
* Substudy inclusion criteria:

  * Completion of the 6-month study period in main study (Visit 10)
  * Randomized and treated with insulin glargine new formulation during the 6-month treatment period (Baseline - month 6)

Exclusion criteria:

* Age less than (<) 18 years
* HbA1c <7.0% or greater than (>) 10% at screening
* Diabetes other than type 2 diabetes mellitus
* Less than 1 year on basal plus mealtime insulin and self-monitoring of blood glucose
* Any contraindication to use of insulin glargine as defined in the national product label
* Participants using human regular insulin as mealtime insulin in the last 3 months before screening visit
* Use of an insulin pump in the last 6 months before screening visit
* Initiation of new glucose-lowering agents and/or weight loss drugs in the last 3 months before screening visit
* History or presence of significant diabetic retinopathy or macular edema likely to require laser or injectable drugs or surgical treatment during the study period
* Pregnant or breast-feeding women or women who intend to become pregnant during the study period
* Substudy exclusion criteria:

  * Participant not willing to use the adaptable injection intervals on at least two days per week

The above information is not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 807 (Actual)
Dates: Start 2011-12; Primary Completion 2013-01 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (193):
- United States (95):
  - Investigational Site Number 840156, Chandler, Arizona
  - Investigational Site Number 840102, Glendale, Arizona
  - Investigational Site Number 840071, Phoenix, Arizona
  - Investigational Site Number 840121, Sun City, Arizona
  - Investigational Site Number 840070, Tempe, Arizona
  - Investigational Site Number 840016, Hot Springs, Arkansas
  - Investigational Site Number 840015, Little Rock, Arkansas
  - Investigational Site Number 840124, Little Rock, Arkansas
  - Investigational Site Number 840032, Searcy, Arkansas
  - Investigational Site Number 840076, Anaheim, California
  - Investigational Site Number 840133, Encino, California
  - Investigational Site Number 840062, Greenbrae, California
  - Investigational Site Number 840057, Huntington Beach, California
  - Investigational Site Number 840059, La Jolla, California
  - Investigational Site Number 840004, La Mesa, California
  - Investigational Site Number 840099, Mission Hills, California
  - Investigational Site Number 840107, Palm Springs, California
  - Investigational Site Number 840005, San Diego, California
  - Investigational Site Number 840013, Tustin, California
  - Investigational Site Number 840002, Walnut Creek, California
  - Investigational Site Number 840114, Colorado Springs, Colorado
  - Investigational Site Number 840136, Colorado Springs, Colorado
  - Investigational Site Number 840092, Longmont, Colorado
  - Investigational Site Number 840049, Daytona Beach, Florida
  - Investigational Site Number 840050, Hollywood, Florida
  - Investigational Site Number 840086, Jacksonville, Florida
  - Investigational Site Number 840011, Jacksonville, Florida
  - Investigational Site Number 840009, Jacksonville, Florida
  - Investigational Site Number 840023, New Port Richey, Florida
  - Investigational Site Number 840012, Ocoee, Florida
  - Investigational Site Number 840148, Palm Harbor, Florida
  - Investigational Site Number 840055, Lawrenceville, Georgia
  - Investigational Site Number 840052, Idaho Falls, Idaho
  - Investigational Site Number 840117, Nampa, Idaho
  - Investigational Site Number 840020, McHenry, Illinois
  - Investigational Site Number 840019, Springfield, Illinois
  - Investigational Site Number 840078, Avon, Indiana
  - Investigational Site Number 840089, Avon, Indiana
  - Investigational Site Number 840097, Avon, Indiana
  - Investigational Site Number 840098, Avon, Indiana
  - Investigational Site Number 840100, Avon, Indiana
  - Investigational Site Number 840127, Vincennes, Indiana
  - Investigational Site Number 840116, Des Moines, Iowa
  - Investigational Site Number 840003, Wichita, Kansas
  - Investigational Site Number 840080, Lexington, Kentucky
  - Investigational Site Number 840042, Paducah, Kentucky
  - Investigational Site Number 840036, Baltimore, Maryland
  - Investigational Site Number 840155, Baltimore, Maryland
  - Investigational Site Number 840034, Rockville, Maryland
  - Investigational Site Number 840065, Ann Arbor, Michigan
  - Investigational Site Number 840066, Dearborn, Michigan
  - Investigational Site Number 840103, Flint, Michigan
  - Investigational Site Number 840126, Kalamazoo, Michigan
  - Investigational Site Number 840022, Southfield, Michigan
  - Investigational Site Number 840143, Chaska, Minnesota
  - Investigational Site Number 840068, Eagan, Minnesota
  - Investigational Site Number 840085, Minneapolis, Minnesota
  - Investigational Site Number 840053, Kalispell, Montana
  - Investigational Site Number 840090, Fremont, Nebraska
  - Investigational Site Number 840091, Omaha, Nebraska
  - Investigational Site Number 840058, Las Vegas, Nevada
  - Investigational Site Number 840043, Brick, New Jersey
  - Investigational Site Number 840152, Toms River, New Jersey
  - Investigational Site Number 840146, Asheville, North Carolina
  - Investigational Site Number 840145, Hickory, North Carolina
  - Investigational Site Number 840045, Wilmington, North Carolina
  - Investigational Site Number 840067, Fargo, North Dakota
  - Investigational Site Number 840008, Cincinnati, Ohio
  - Investigational Site Number 840106, Columbus, Ohio
  - Investigational Site Number 840123, Dayton, Ohio
  - Investigational Site Number 840119, Maumee, Ohio
  - Investigational Site Number 840122, Mentor, Ohio
  - Investigational Site Number 840083, Medford, Oregon
  - Investigational Site Number 840084, Portland, Oregon
  - Investigational Site Number 840007, Uniontown, Pennsylvania
  - Investigational Site Number 840079, Greer, South Carolina
  - Investigational Site Number 840048, Rapid City, South Dakota
  - Investigational Site Number 840039, Chattanooga, Tennessee
  - Investigational Site Number 840159, Knoxville, Tennessee
  - Investigational Site Number 840021, Austin, Texas
  - Investigational Site Number 840129, Austin, Texas
  - Investigational Site Number 840081, Austin, Texas
  - Investigational Site Number 840001, Dallas, Texas
  - Investigational Site Number 840047, Dallas, Texas
  - Investigational Site Number 840082, Houston, Texas
  - Investigational Site Number 840120, Hurst, Texas
  - Investigational Site Number 840010, Draper, Utah
  - Investigational Site Number 840060, Ogden, Utah
  - Investigational Site Number 840035, Chesapeake, Virginia
  - Investigational Site Number 840074, Norfolk, Virginia
  - Investigational Site Number 840112, Norfolk, Virginia
  - Investigational Site Number 840041, Norfolk, Virginia
  - Investigational Site Number 840104, Richmond, Virginia
  - Investigational Site Number 840075, Williamsburg, Virginia
  - Investigational Site Number 840018, Milwaukee, Wisconsin
- Canada (22):
  - Investigational Site Number 124024, Beamsville
  - Investigational Site Number 124025, Burlington
  - Investigational Site Number 124023, Calgary
  - Investigational Site Number 124020, Calgary
  - Investigational Site Number 124019, Chatham
  - Investigational Site Number 124018, Coquitlam
  - Investigational Site Number 124021, Hamilton
  - Investigational Site Number 124014, Hamilton
  - Investigational Site Number 124006, Laval
  - Investigational Site Number 124009, London
  - Investigational Site Number 124008, Mississauga
  - Investigational Site Number 124015, Montreal
  - Investigational Site Number 124004, Montreal
  - Investigational Site Number 124005, Oshawa
  - Investigational Site Number 124026, Québec
  - Investigational Site Number 124002, Red Deer
  - Investigational Site Number 124017, Saint-Laurent
  - Investigational Site Number 124007, Thornhill
  - Investigational Site Number 124001, Toronto
  - Investigational Site Number 124011, Toronto
  - Investigational Site Number 124010, Victoria
  - Investigational Site Number 124022, Winnipeg
- Czechia (10):
  - Investigational Site Number 203006, Beroun
  - Investigational Site Number 203001, Břeclav
  - Investigational Site Number 203002, Hodonín
  - Investigational Site Number 203009, Holešov
  - Investigational Site Number 203003, Hradec Králové
  - Investigational Site Number 203007, Hranice
  - Investigational Site Number 203004, Krnov
  - Investigational Site Number 203010, Olomouc
  - Investigational Site Number 203008, Prague
  - Investigational Site Number 203005, Prostějov
- Estonia (6):
  - Investigational Site Number 233002, Pärnu
  - Investigational Site Number 233004, Tallinn
  - Investigational Site Number 233006, Tallinn
  - Investigational Site Number 233003, Tallinn
  - Investigational Site Number 233001, Tallinn
  - Investigational Site Number 233005, Tartu
- Finland (3):
  - Investigational Site Number 246001, Helsinki
  - Investigational Site Number 246005, Kuopio
  - Investigational Site Number 246002, Oulu
- France (2):
  - Investigational Site Number 250004, La Rochelle
  - Investigational Site Number 250002, Strasbourg
- Germany (3):
  - Investigational Site Number 276006, Heidelberg
  - Investigational Site Number 276002, Riesa
  - Investigational Site Number 276003, Schwabenheim
- Hungary (17):
  - Investigational Site Number 348010, Baja
  - Investigational Site Number 348004, Balatonfüred
  - Investigational Site Number 348015, Budapest
  - Investigational Site Number 348013, Budapest
  - Investigational Site Number 348017, Budapest
  - Investigational Site Number 348009, Budapest
  - Investigational Site Number 348002, Budapest
  - Investigational Site Number 348005, Debrecen
  - Investigational Site Number 348008, Eger
  - Investigational Site Number 348018, Gyula
  - Investigational Site Number 348014, Makó
  - Investigational Site Number 348012, Mosonmagyaróvár
  - Investigational Site Number 348007, Nyiregyháza
  - Investigational Site Number 348011, Sátorlaljaújhely
  - Investigational Site Number 348003, Szeged
  - Investigational Site Number 348006, Szombathely
  - Investigational Site Number 348001, Zalaegerszeg
- Latvia (6):
  - Investigational Site Number 428006, Jēkabpils
  - Investigational Site Number 428005, Ogre
  - Investigational Site Number 428002, Riga
  - Investigational Site Number 428001, Riga
  - Investigational Site Number 428004, Riga
  - Investigational Site Number 428003, Sigulda
- Mexico (5):
  - Investigational Site Number 484007, Chihuahua City
  - Investigational Site Number 484001, Cuernavaca
  - Investigational Site Number 484006, Guadalajara
  - Investigational Site Number 484003, Monterrey
  - Investigational Site Number 484004, Pachuca
- Netherlands (8):
  - Investigational Site Number 528009, Almelo
  - Investigational Site Number 528004, Eindhoven
  - Investigational Site Number 528007, Groningen
  - Investigational Site Number 528005, Hoogeveen
  - Investigational Site Number 528001, Hoorn
  - Investigational Site Number 528008, Leeuwarden
  - Investigational Site Number 528006, Utrecht
  - Investigational Site Number 528002, Venlo
- Romania (9):
  - Investigational Site Number 642001, Bacau
  - Investigational Site Number 642005, Bucharest
  - Investigational Site Number 642006, Bucharest
  - Investigational Site Number 642002, Cluj-Napoca
  - Investigational Site Number 642004, Iași
  - Investigational Site Number 642008, Iași
  - Investigational Site Number 642003, Oradea
  - Investigational Site Number 642009, Târgu Mureş
  - Investigational Site Number 642007, Timișoara
- South Africa (7):
  - Investigational Site Number 710005, Alberton
  - Investigational Site Number 710003, Johannesburg
  - Investigational Site Number 710006, Lenasia
  - Investigational Site Number 710002, Observatory
  - Investigational Site Number 710001, Paarl
  - Investigational Site Number 710008, Pretoria
  - Investigational Site Number 710004, Somerset West

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Result] Riddle MC, Bolli GB, Ziemen M, Muehlen-Bartmer I, Bizet F, Home PD; EDITION 1 Study Investigators. New insulin glargine 300 units/mL versus glargine 100 units/mL in people with type 2 diabetes using basal and mealtime insulin: glucose control and hypoglycemia in a 6-month randomized controlled trial (EDITION 1). Diabetes Care. 2014 Oct;37(10):2755-62. doi: 10.2337/dc14-0991. Epub 2014 Jul 30. PMID 25078900
- [Derived] Yale JF, Aroda VR, Charbonnel B, Sinclair AJ, Trescoli C, Cahn A, Bigot G, Merino-Trigo A, Brulle-Wohlhueter C, Bolli GB, Ritzel R. Glycaemic control and hypoglycaemia risk with insulin glargine 300 U/mL versus glargine 100 U/mL: A patient-level meta-analysis examining older and younger adults with type 2 diabetes. Diabetes Metab. 2020 Apr;46(2):110-118. doi: 10.1016/j.diabet.2018.10.002. Epub 2018 Oct 23. PMID 30366067
- [Derived] Bonadonna RC, Renard E, Cheng A, Fritsche A, Cali A, Melas-Melt L, Umpierrez GE. Switching to insulin glargine 300 U/mL: Is duration of prior basal insulin therapy important? Diabetes Res Clin Pract. 2018 Aug;142:19-25. doi: 10.1016/j.diabres.2018.03.041. Epub 2018 Apr 9. PMID 29649539

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 1177 participants were screened, of whom 370 participants were screen failure and 807 participants were randomized.
Pre-assignment Details: Following the main 6 month treatment period, eligible participants previously using HOE901-U300 were randomized (1:1) in a substudy and continued with fixed-dosing (every 24 hours) or started a adaptable-dosing (at intervals of 24 +/- 3 hours) regimen for 3 Months (Month 6 to 9).
Groups:
- HOE901-U300: HOE901-U300 (new insulin glargine 300 units per milliliter [U/mL]) subcutaneous (SC) injection once daily (evening) for 12 months on top of mealtime insulin analogue.
- Lantus: Lantus (HOE901-U100, insulin glargine 100 U/mL) SC injection once daily (evening) for 12 months on top of mealtime insulin analogue.
Period: Overall Study
Arm/Group | HOE901-U300 | Lantus
Started | 404 | 403
Treated | 404 | 402
Participated in Substudy | 109 (56 participants received adaptable dosing regimen and 53 participants received fixed dosing regimen) | 0
Modified Intent-to-Treat Population | 404 (Participants who received at least 1 dose of drug, had both baseline, at least 1 post-baseline data) | 400 (Participants who received at least 1 dose of drug, had both baseline, at least 1 post-baseline data)
Completed | 359 | 355
Not Completed | 45 | 48
Not completed — Randomized but not Treated | 0 | 1
Not completed — Adverse Event | 12 | 16
Not completed — Lack of Efficacy | 1 | 1
Not completed — Protocol Violation | 6 | 8
Not completed — Diverse Reasons | 18 | 14
Not completed — Site Closure for Noncompliance | 5 | 2
Not completed — Hypoglycemia | 2 | 3
Not completed — Lost to Follow-up | 1 | 3

BASELINE CHARACTERISTICS:
Population: Randomized population: all screened participants (who originally met inclusion criteria and signed informed consent) allocated to a treatment group and recorded in Interactive Voice/Web Response System (IVRS/IWRS) database, regardless of whether treatment was used or not. Participants were analyzed in treatment group to which they were randomized.
Groups:
- HOE901-U300: HOE901-U300 SC injection once daily for 12 months on top of mealtime insulin.
- Lantus: Lantus SC injection once daily for 12 months on top of mealtime insulin.
- Total: Total of all reporting groups
Arm/Group | HOE901-U300 | Lantus | Total
Number analyzed (Participants) | 404 | 403 | 807
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.1 (8.5) | 59.8 (8.7) | 60.0 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 187 | 193 | 380
  Male | 217 | 210 | 427
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)] | 36.6 (6.8) | 36.6 (6.1) | 36.6 (6.4)
Duration of Diabetes [Mean (Standard Deviation); unit: years] | 15.6 (7.2) | 16.1 (7.8) | 15.8 (7.5)
Basal Insulin Daily Dose [Mean (Standard Deviation); unit: units per kilogram (U/kg)] — Number of participants analyzed for this baseline characteristics = 372 and 361 in HOE901-U300 and Lantus arm, respectively.
  units per kilogram (U/kg) | 0.668 (0.263) | 0.667 (0.241) | 0.668 (0.252)
Total Insulin Daily Dose [Mean (Standard Deviation); unit: U/kg] — Number of participants analyzed for this baseline characteristics = 367 and 360 in HOE901-U300 and Lantus arm, respectively
  U/kg | 1.194 (0.483) | 1.200 (0.448) | 1.197 (0.466)
Glycated Hemoglobin A1c (HbA1c) [Number; unit: participants]
  Less Than (<) 8% | 144 | 144 | 288
  Greater Than or Equal to (>=) 8% | 260 | 259 | 519

OUTCOME MEASURES:

1. Primary Outcome: Change in HbA1c From Baseline to Month 6 Endpoint
Time Frame: Baseline, Month 6
Population: Modified Intent-to-Treat population: all randomized participants who received at least (>=)1 dose, had baseline and >=1 post-baseline assessment of any efficacy variable, irrespective of compliance. Number of participants analyzed = participants with baseline and Week 6 HbA1c assessment. Missing data imputed using last observation carried forward.
Measure: Least Squares Mean (Standard Error); unit: percentage of hemoglobin
Arm/Group | HOE901-U300 | Lantus
Number analyzed (Participants) | 391 | 394
percentage of hemoglobin | -0.83 (0.060) | -0.83 (0.061)
Statistical Analysis 1: Comparison: HOE901-U300 vs Lantus; Analysis was performed using an analysis of covariance (ANCOVA) model with treatment, strata of screening HbA1c (<8.0 and >=8.0%), and country as fixed effects and using the HbA1c baseline value as a covariate; Test type: Non-Inferiority or Equivalence — Stepwise closed testing approach was used to assess non-inferiority and superiority sequentially: 1. Non-inferiority of HOE901-U300 vs Lantus: Upper bound of two-sided 95% confidence interval (CI) of difference between HOE901-U300 and Lantus on mITT population is <0.4%. 2. Superiority (only if non-inferiority has been demonstrated): Upper bound of two-sided 95% CI for difference in mean change in HbA1c from baseline to endpoint between HOE901-U300 and Lantus on mITT population is <0; Least Squares (LS) Mean Difference = -0.00, 95% CI 2-sided [-0.112 to 0.107], Standard Error of Mean 0.056

2. Secondary Outcome: Percentage of Participants With At Least One Severe and/or Confirmed Nocturnal Hypoglycemia From Start of Week 9 to Month 6 Endpoint
Description: Nocturnal hypoglycemia was hypoglycemia that occurred between 00:00 and 05:59 hours (clock time), regardless the participant was awake or woke up because of the event. Severe hypoglycemia was an event that required assistance of another person to actively administer carbohydrate, glucagon, or other resuscitative actions. Confirmed hypoglycemia was an event associated with plasma glucose less than or equal to (<=) 3.9 millimoles per liter (mmol/L) (70 milligram per deciliter [mg/dL]).
Time Frame: Week 9 Up to Month 6
Population: Modified intent-to-treat population.
Measure: Number; unit: percentage of participants
Arm/Group | HOE901-U300 | Lantus
Number analyzed (Participants) | 404 | 400
percentage of participants | 36.1 | 46.0
Statistical Analysis 1: Comparison: HOE901-U300 vs Lantus; A one-sided test (at alpha=0.025) for superiority of HOE901-U300 over Lantus was to be performed in case the non-inferiority of HOE901-U300 vs Lantus for the primary endpoint was demonstrated. Analysis was performed using Cochran-Mantel-Haenszel (CMH) method with treatment as a factor and stratified on strata of screening HbA1c (<8.0 and >=8.0%); Test type: Superiority or Other; p = 0.0045, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 0.79, 95% CI 2-sided [0.67 to 0.93]

3. Secondary Outcome: Change in Average Preinjection Self-Monitored Plasma Glucose (SMPG) From Baseline to Month 6 Endpoint
Description: Pre-injection SMPG was measured within 30 minutes prior to the injection of the study drug. Average was assessed by the mean of at least 3 SMPG calculated over the 7 days preceding the assessment visit.
Time Frame: Baseline, Month 6
Population: mITT population. Missing data imputed using last observation carried forward. Number of participants analyzed = participants with baseline and Month 6 pre-injection SMPG assessment.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | HOE901-U300 | Lantus
Number analyzed (Participants) | 365 | 360
mmol/L | -0.90 (0.182) | -0.84 (0.182)
Statistical Analysis 1: Comparison: HOE901-U300 vs Lantus; Change in pre-injection SMPG was analyzed using an ANCOVA model with treatment, strata of screening HbA1c (<8.0 and >=8.0%), and country as fixed effects and using the pre-injection SMPG baseline value as a covariate. A test for superiority of HOE901-U300 over Lantus was to be performed one-sided at level alpha = 0.025 if previous analysis for nocturnal hypoglycemia was significant; Test type: Superiority or Other; p = 0.6909, ANCOVA; LS Mean Difference = -0.06, 95% CI 2-sided [-0.383 to 0.254], Standard Error of Mean 0.162

4. Secondary Outcome: Change in Variability of Preinjection SMPG From Baseline to Month 6 Endpoint
Description: Pre-injection SMPG was measured within 30 minutes prior to the injection of the study drug. Variability was assessed by the mean of coefficient of variation calculated as 100 multiplied by (standard deviation/mean) over at least 3 SMPG measured during the 7 days preceding the assessment visit.
Time Frame: Baseline, Month 6
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: percentage of mean
Arm/Group | HOE901-U300 | Lantus
Number analyzed (Participants) | 365 | 360
percentage of mean | -1.10 (1.222) | -1.08 (1.222)

5. Secondary Outcome: Percentage of Participants With HbA1c <7% at Month 6 Endpoint
Time Frame: Month 6
Population: mITT Population. Number of participants analyzed = participants with baseline and Month 6 HbA1c assessment. Missing data imputed using last observation carried forward.
Measure: Number; unit: percentage of participants
Arm/Group | HOE901-U300 | Lantus
Number analyzed (Participants) | 391 | 394
percentage of participants | 39.6 | 40.9

6. Secondary Outcome: Change in Fasting Plasma Glucose (FPG) From Baseline to Month 6 Endpoint
Time Frame: Baseline, Month 6
Population: mITT Population. Number of participants analyzed = participants with baseline and Month 6 FPG assessment. Missing data imputed using last observation carried forward.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | HOE901-U300 | Lantus
Number analyzed (Participants) | 376 | 385
mmol/L | -1.29 (0.191) | -1.38 (0.192)

7. Secondary Outcome: Percentage of Participants With FPG <5.6 mmol/L (<100 mg/dL) at Month 6 Endpoint
Time Frame: Month 6
Population: mITT Population. Number of participants analyzed = participants with Month 6 FPG assessment. Missing data imputed using last observation carried forward.
Measure: Number; unit: percentage of participants
Arm/Group | HOE901-U300 | Lantus
Number analyzed (Participants) | 389 | 392
percentage of participants | 26.5 | 23.2

8. Secondary Outcome: Change in 8-Point SMPG Profiles Per Time Point From Baseline to Month 6 Endpoint
Description: Change in each time-point of 8-point SMPG profile: 03:00 hours (clock time) at night; before and 2 hours after breakfast; before and 2 hours after lunch; before and 2 hours after dinner; and at bedtime.
Time Frame: Baseline, Month 6
Population: mITT Population. Here, n = participants with Baseline and Month 6 8-point SMPG assessment separately for each analysed time point. Missing data imputed using last observation carried forward.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | HOE901-U300 | Lantus
Number analyzed (Participants) | 404 | 400
mmol/L
  03:00 at Night Plasma Glucose (n=333,323) | -0.98 (0.248) | -1.16 (0.251)
  Pre-Breakfast Plasma Glucose (n=343,333) | -1.19 (0.189) | -1.49 (0.190)
  2 Hours After Breakfast Plasma Glucose (n=335,326) | -1.60 (0.241) | -1.90 (0.243)
  Pre-Lunch Plasma Glucose (n=337,331) | -1.05 (0.213) | -1.23 (0.216)
  2 Hours After Lunch Plasma Glucose (n=336,325) | -0.64 (0.280) | -0.63 (0.282)
  Pre-Dinner Plasma Glucose (n=338,333) | -0.47 (0.261) | -0.37 (0.260)
  2 Hours After Dinner Plasma Glucose (n=331,327) | -0.96 (0.298) | -1.17 (0.298)
  Bedtime Plasma Glucose (n=324, 325) | -0.88 (0.324) | -0.91 (0.326)

9. Secondary Outcome: Change in Daily Basal Insulin Dose From Baseline to Month 6 Endpoint
Time Frame: Baseline, Month 6
Population: mITT Population. Number of participants analyzed = participants with Baseline and Month 6 basal insulin dose assessment. Missing data imputed using last observation carried forward.
Measure: Least Squares Mean (Standard Error); unit: U/kg
Arm/Group | HOE901-U300 | Lantus
Number analyzed (Participants) | 403 | 400
U/kg | 0.28 (0.017) | 0.19 (0.017)

10. Secondary Outcome: Change in Treatment Satisfaction Score Using The Diabetes Treatment Satisfaction Questionnaire (DTSQs) From Baseline to Month 6 Endpoint
Description: DTSQ is a validated measure to assess how satisfied participants with diabetes are with their treatment and how they perceive hyper- and hypoglycemia. It consists of 8 questions which are answered on a Likert scale from 0 to 6. DTSQ treatment satisfaction score is the sum of question 1 and 4-8 scores and ranges between 0 and 36, where higher scores indicate more treatment satisfaction.
Time Frame: Baseline, Month 6
Population: mITT Population. Number of participants analyzed = participants with Baseline and Month 6 DTSQ assessment. Missing data imputed using last observation carried forward.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | HOE901-U300 | Lantus
Number analyzed (Participants) | 366 | 363
units on a scale | 2.32 (0.310) | 2.24 (0.313)

11. Secondary Outcome: Percentage of Participants With Hypoglycemia (All and Nocturnal) Events From Baseline up to Month 12
Description: Hypoglycemia events were Severe hypoglycemia (an event that required assistance of another person to actively administer carbohydrate, glucagon, or other resuscitative actions); Documented symptomatic hypoglycemia (typical symptoms of hypoglycemia with plasma glucose level of <=3.9 mmol/L [70 mg/dL]); Asymptomatic hypoglycemia (no typical symptoms of hypoglycemia but plasma glucose level <=3.9 mmol/L); Probable symptomatic hypoglycemia (an event during which symptoms of hypoglycemia were not accompanied by a plasma glucose determination, but was presumably caused by a plasma glucose level <=3.9 mmol/L, symptoms treated with oral carbohydrate without a test of plasma glucose); Relative hypoglycemia (an event during which the person with diabetes reported any of the typical symptoms of hypoglycemia, and interpreted the symptoms as indicative of hypoglycemia, but plasma glucose level >3.9 mmol/L); Severe and/or confirmed a hypoglycemia (plasma glucose <=3.9 mmol/L).
Time Frame: Up to Month 12
Population: Safety population: all participants randomized and exposed to at least one dose of study drug, regardless of the amount of treatment administered. In the event of participants having received treatments different from those assigned according to the randomization schedule, safety analyses were conducted according to treatment received.
Measure: Number; unit: percentage of participants
Arm/Group | HOE901-U300 | Lantus
Number analyzed (Participants) | 404 | 402
percentage of participants
  Any Hypoglycemia Event: All Hypoglycemia | 87.4 | 92.0
  Severe Hypoglycemia: All Hypoglycemia | 6.7 | 7.5
  Documented Symptomatic: All Hypoglycemia | 74.8 | 82.8
  Asymptomatic: All Hypoglycemia | 70.5 | 73.4
  Probable Symptomatic: All Hypoglycemia | 5.7 | 8.5
  Relative: All Hypoglycemia | 15.8 | 21.1
  Severe and/or Confirmed: All Hypoglycemia | 85.9 | 91.5
  Any Hypoglycemia Event: Nocturnal Hypoglycemia | 55.4 | 66.2
  Severe Hypoglycemia: Nocturnal | 2.5 | 3.2
  Documented Symptomatic: Nocturnal Hypoglycemia | 44.6 | 57.2
  Asymptomatic: Nocturnal Hypoglycemia | 29.2 | 31.1
  Probable Symptomatic: Nocturnal Hypoglycemia | 2.2 | 2.7
  Relative: Nocturnal Hypoglycemia | 5.0 | 10.0
  Severe and/or Confirmed: Nocturnal Hypoglycemia | 54.5 | 64.7

12. Other Pre Specified Outcome: Change in HbA1c From Month 6 to Month 9
Description: Substudy comparing fixed dosing regimen (every 24 hours) vs. adaptive dosing regimen (every 24 +/- 3 hours) in a subset of participants randomized to HOE901-U300 and treated for 6 months.
Time Frame: Month 6 Up to Month 9
Population: mITT substudy population. Number of participants analyzed = participants with Month 6 and Month 9 HbA1c assessment. Analysis was planned to be performed for participants enrolled in the substudy and who were receiving HOE901-U300 (Adaptable dosing intervals or Fixed dosing intervals).
Measure: Least Squares Mean (Standard Error); unit: percentage of hemoglobin
Groups:
- HOE901-U300: Adaptable Dosing Intervals: HOE901-U300 SC injection once daily for 6 months on top of mealtime insulin. From Month 6 to Month 9 participants received HOE901-U300 once daily at intervals of 24 +/- 3 hours.
- HOE901-U300: Fixed Dosing Intervals: HOE901-U300 SC injection once daily for 6 months on top of mealtime insulin. From Month 6 up to Month 9 participants received HOE901-U300 once daily every 24 hours.
Arm/Group | HOE901-U300: Adaptable Dosing Intervals | HOE901-U300: Fixed Dosing Intervals
Number analyzed (Participants) | 55 | 51
percentage of hemoglobin | 0.21 (0.111) | 0.15 (0.120)
Statistical Analysis 1: Comparison: HOE901-U300: Adaptable Dosing Intervals vs HOE901-U300: Fixed Dosing Intervals; Analysis was performed using Analysis of covariance (ANCOVA) model with treatment regimen and country as fixed effects and baseline HbA1c value as a covariate; Test type: Superiority or Other; LS Mean Difference = 0.05, 95% CI 2-sided [-0.189 to 0.298], Standard Error of Mean 0.123

ADVERSE EVENTS:
Time Frame: All Adverse Events (AE) were collected from signature of the informed consent form up to 12 months regardless of seriousness or relationship to investigational product.
Description: Reported adverse events are treatment-emergent adverse events that is AEs that developed/worsened during the 'on treatment period' (time from the first injection of study drug up to 2 days (1 day for FPG, SMPG; 0 day for insulin glargine dose) after the last injection of study drug). Analysis was done on safety population.
Arm/Group | HOE901-U300 | Lantus
Serious Adverse Events (participants affected / at risk) | 53/404 | 62/402
Other Adverse Events (participants affected / at risk) | 131/404 | 132/402
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HOE901-U300 (N=404) | Lantus (N=402)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 0 | 2
Angina unstable (Cardiac disorders) | 0 | 1
Aortic valve stenosis (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 2 | 3
Bundle branch block left (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 1 | 1
Cardiac failure chronic (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 1
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 3 | 1
Myocardial infarction (Cardiac disorders) | 1 | 1
Myocardial ischaemia (Cardiac disorders) | 1 | 1
Palpitations (Cardiac disorders) | 1 | 0
Pulseless electrical activity (Cardiac disorders) | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1
Diverticulitis intestinal haemorrhagic (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 1 | 1
Non-cardiac chest pain (General disorders) | 1 | 1
Bile duct stone (Hepatobiliary disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Anaphylactic reaction (Immune system disorders) | 0 | 1
Bronchitis (Infections and infestations) | 2 | 0
Bronchopneumonia (Infections and infestations) | 2 | 0
Cellulitis (Infections and infestations) | 3 | 1
Diverticulitis (Infections and infestations) | 0 | 1
Endocarditis (Infections and infestations) | 1 | 0
Erysipelas (Infections and infestations) | 1 | 1
Gastroenteritis (Infections and infestations) | 0 | 2
Groin abscess (Infections and infestations) | 1 | 0
Infected skin ulcer (Infections and infestations) | 1 | 0
Lyme disease (Infections and infestations) | 0 | 1
Osteomyelitis (Infections and infestations) | 3 | 2
Pneumonia (Infections and infestations) | 0 | 3
Pneumonia mycoplasmal (Infections and infestations) | 0 | 1
Postoperative wound infection (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 1
Pyelonephritis acute (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 1 | 1
Septic embolus (Infections and infestations) | 1 | 0
Tracheobronchitis (Infections and infestations) | 0 | 1
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0
Airway complication of anaesthesia (Injury, poisoning and procedural complications) | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 2 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 2
Lactose intolerance (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 2 | 0
Spondylitis (Musculoskeletal and connective tissue disorders) | 1 | 1
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 | 1
B-cell small lymphocytic lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast angiosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Meningioma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Altered state of consciousness (Nervous system disorders) | 0 | 1
Cerebral infarction (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Cervicobrachial syndrome (Nervous system disorders) | 0 | 1
Guillain-Barre syndrome (Nervous system disorders) | 0 | 1
Hypoglycaemic unconsciousness (Nervous system disorders) | 2 | 0
Syncope (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 1
Depression (Psychiatric disorders) | 0 | 1
Diabetic nephropathy (Renal and urinary disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 1
Renal failure chronic (Renal and urinary disorders) | 0 | 3
Urinary bladder polyp (Renal and urinary disorders) | 1 | 0
Metrorrhagia (Reproductive system and breast disorders) | 1 | 0
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 1 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 | 1
Skin ulcer haemorrhage (Skin and subcutaneous tissue disorders) | 0 | 1
Accelerated hypertension (Vascular disorders) | 0 | 1
Aortic stenosis (Vascular disorders) | 0 | 1
Extremity necrosis (Vascular disorders) | 0 | 1
Intermittent claudication (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | HOE901-U300 (N=404) | Lantus (N=402)
Diarrhoea (Gastrointestinal disorders) | 22 | 21
Bronchitis (Infections and infestations) | 23 | 30
Influenza (Infections and infestations) | 22 | 18
Nasopharyngitis (Infections and infestations) | 34 | 36
Sinusitis (Infections and infestations) | 21 | 15
Upper respiratory tract infection (Infections and infestations) | 38 | 34
Arthralgia (Musculoskeletal and connective tissue disorders) | 13 | 21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.